CLINICAL TRIAL: NCT00808574
Title: Effect of a Web-Based Presentation on Communication With Healthcare Providers
Brief Title: Screening for Obstructive Sleep Apnea Among Members of an Internet Weight Loss Community
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Kevin O. Hwang, M.D., M.P.H. (principle investigator), The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: HSC-MS-08-0346
Record Dates: First submitted 2008-12-12; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Internet; Screening; Health belief model
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Brief, theory-based, online assessment of OSA risk followed by risk-tailed OSA presentation.
  Interventions: Behavioral: Obstructive sleep apnea screening intervention
- Control (No Intervention): No risk assessment or presentation

INTERVENTIONS:
Behavioral: Obstructive sleep apnea screening intervention — Brief, theory-based, online assessment of OSA risk followed by risk-tailed OSA presentation.
  Arms: Intervention

SUMMARY:
The current study was a pilot, double blind, randomized controlled trial to (1) evaluate the feasibility of an online obstructive sleep apnea (OSA) screening intervention, (2) estimate effect size for planning of future studies, and (3) test the hypothesis that the intervention, compared to a control condition, would lead more individuals to discuss OSA with their healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* Member of SparkPeople.com community and logged on within previous month
* Live in the US

Exclusion Criteria:

* Prior diagnosis of OSA
* Prior discussions with healthcare provider about OSA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Online questionnaire asking whether subject has discussed OSA with healthcare provider since enrolling in study | 12 weeks

SECONDARY OUTCOMES:
Online questionnaire asking whether subject has plans to discuss OSA with healthcare provider, if not done already | 12 weeks
Online questionnaire asking whether subject has undergone testing and treatment for OSA since enrolling in study | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O Hwang, MD, MPH, Principal Investigator — University of Texas Medical School, Houston
Locations (1):
- University of Texas Medical School, Houston, Houston, Texas, United States